CLINICAL TRIAL: NCT00486993
Title: Estimation of Prevalence and Assessment of the Effects of Modification of Cardiovascular Risk Factors in an Ambulatory Urban Patient Population
Brief Title: Cardiovascular Risk Factors in an Ambulatory Urban Patient Population
Acronym: AsuRiesgo
Status: Completed | Type: Observational
Sponsor: Heidelberg University (Other)
Responsible Party: Principal Investigator, Derliz Mereles, Head Echocardiography Laboratory, Heidelberg University
Other Study IDs: AsuRiesgo
Record Dates: First submitted 2007-06-12; First posted 2007-06-15 (Estimated); Last update posted 2016-11-08 (Estimated); Status verified 2016-11

CONDITIONS: Cardiovascular Risk Factors; Metabolic Syndrome; Lifestyle Modification; Coronary Artery Disease; Stroke
Keywords: Diet; Exercise; Smoking; Stress; Polyphenols
MeSH Terms: conditions — Metabolic Syndrome; Coronary Artery Disease; Stroke; Motor Activity; Smoking | interventions — Diet

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- asuriesgo: unselected outpatient population
  Interventions: Behavioral: Dietary and nutritional modification; Behavioral: Stop smoking; Behavioral: Regular physical activities; Behavioral: Weight reduction to normal ranges; Behavioral: Regular intake of polyphenols, esp. from Ilex paraguayensis

INTERVENTIONS:
Behavioral: Dietary and nutritional modification
Behavioral: Stop smoking
Behavioral: Regular physical activities
Behavioral: Weight reduction to normal ranges
Behavioral: Regular intake of polyphenols, esp. from Ilex paraguayensis

SUMMARY:
According to WHO estimations, cardiovascular diseases (CVDs) are the number one cause of death globally. More people die annually from CVDs than from any other cause. An estimated 17.5 million people died from CVDs in 2005, representing 30% of all global deaths. Of these deaths, an estimated 7.6 million were due to coronary heart disease and 5.7 million were due to stroke.

Over 80% of CVD deaths take place in low- and middle-income countries and occur almost equally in men and women. In Paraguay, prevalence of classic risk factors, as well as new ones, like the metabolic syndrome are not completely known.

Government health policies in industrialized countries are focusing on programs to modify cardiovascular risk factors. In developing countries, prevention of coronary heart disease and stroke through modification of cardiovascular risk factors are not playing a large role at the moment.

The aim of this study is to define the effects of changes in lifestyle on cardiovascular risk factors, when added to optimized standard pharmacological therapy for arterial hypertension, diabetes mellitus and hyperlipidemia, in an ambulatory urban patient population.

ELIGIBILITY:
Inclusion Criteria:

* all ambulatory patients, with age 18 years or older

Exclusion Criteria:

* no exclusion criteria provided, particularly for the first, epidemiological part of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: unselected outpatient population
Sampling Method: Non-Probability Sample
Enrollment: 18287 (Actual)
Dates: Start 2006-05; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
cardiovascular mortality | one year

SECONDARY OUTCOMES:
mortality, other causes | one year
acute myocardial infarction | one year
stroke | one year
acute coronary syndrome | one year

CONTACTS AND LOCATIONS:
Overall Officials: Derliz Mereles, MD, Principal Investigator — Heidelberg University
Locations (1):
- Hospital Central Instituto de Prevision Social, Asunción, Dep. Central, Paraguay

REFERENCES:
- [Background] Jimenez JT, Palacios M, Canete F, Barriocanal LA, Medina U, Figueredo R, Martinez S, de Melgarejo MV, Weik S, Kiefer R, Alberti KG, Moreno-Azorero R. Prevalence of diabetes mellitus and associated cardiovascular risk factors in an adult urban population in Paraguay. Diabet Med. 1998 Apr;15(4):334-8. doi: 10.1002/(SICI)1096-9136(199804)15:43.0.CO;2-Z. PMID 9585400
- [Background] Ramirez MO, Pino CT, Furiasse LV, Lee AJ, Fowkes FG. Paraguayan National Blood Pressure Study: prevalence of hypertension in the general population. J Hum Hypertens. 1995 Nov;9(11):891-7. PMID 8583468
- See also: Internet site of the study — http://www.asuriesgo.de